CLINICAL TRIAL: NCT00111735
Title: What is the Optimal Serum TSH Concentration During Thyroxine Treatment for Primary Hypothyroidism? Effects of Fine Titration of Thyroxine Dosage on Wellbeing, Quality of Life and Cognitive Function
Brief Title: Thyroxine Titration Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sir Charles Gairdner Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2003-015
Record Dates: First submitted 2005-05-24; First posted 2005-05-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-05

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroxine

INTERVENTIONS:
Drug: Thyroxine

SUMMARY:
The aim of the study is to examine the effects of fine titration of thyroxine dosage on symptoms of hypothyroidism, wellbeing and quality of life. The hypothesis is that symptoms of hypothyroidism, wellbeing and quality of life will be improved in thyroxine-treated subjects when serum thyrotropin (TSH) is suppressed and/or in the lower reference range, compared to when TSH is in the upper reference range.

DETAILED DESCRIPTION:
Primary hypothyroidism is a common disorder, affecting 2% of the Australian population. The standard treatment is with thyroxine (T4), and conventionally, a serum thyrotropin (TSH) concentration within the laboratory range is taken as indicating adequacy of thyroxine dosage.

Some patients with hypothyroidism complain of persistently impaired well-being, despite taking thyroxine in a dose which normalises serum TSH concentrations. It is not clear whether this is because of comorbidity or because standard thyroxine replacement is in some way inadequate for some individuals.

The reference range for serum TSH is wide (currently 0.34-4.8 mU/L at PathCentre). The distribution of serum TSH concentrations in the population is skewed, with the mean and median in the lower reference range at approximately 1.0 mU/L. This has led some to argue that a serum TSH in the lower reference range should be the usual therapeutic target. Anecdotal evidence suggests that some thyroxine-treated patients do feel better if the thyroxine dose is adjusted so that serum TSH is in the lower reference range rather than the upper reference range. The National Academy for Clinical Biochemistry of the United States now recommends, that for thyroxine-treated patients, that serum TSH should be less than 2.0 mU/L. There is, however, no evidence from properly conducted studies that aiming for a serum TSH concentration in the lower reference range improves symptoms of hypothyroidism or general wellbeing, and this proposal has not been generally adopted.

Only one study examining the effects of fine titration of thyroxine dosage on wellbeing has been published. In this study, patients had significantly improved wellbeing if they took a dose of thyroxine which was 50 μg greater than their biochemically optimal dose as determined by a thyrotropin-releasing hormone test. In most cases, serum TSH was suppressed to below 0.2 mU/L (the limit of sensitivity of the assay) on the thyroxine doses which improved wellbeing. This study was open-label and non-randomised, and the results therefore may have been affected by bias.

A well-designed, double blind study of the effects of fine titration of thyroxine dosage on symptoms of hypothyroidism, wellbeing and quality of life is required to determine if a serum TSH in the lower reference range, rather than simply TSH within the reference range, should indeed be the usual therapeutic target for thyroxine therapy in primary hypothyroidism. It is also desirable to confirm the findings of Carr et al., that patients have improved wellbeing if TSH is suppressed to below normal levels.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects >18 years of age
* Primary hypothyroidism ≥6 months duration arising from autoimmune hypothyroidism, thyroidectomy or radioiodine treatment
* Thyroxine dose ≥100 mcg/day
* No change in thyroxine dose in past 2 months
* Serum TSH of 0.1-4.8 mU/L
* Adequate contraceptive measures for women of childbearing age

Exclusion Criteria:

* Major systemic illness affecting quality of life or likely to affect participation in the study
* Treatment with T3 currently or in past 2 months
* History of thyroid cancer requiring suppression of TSH secretion by thyroxine
* Ischaemic heart disease - previous myocardial infarction, angina or coronary artery revascularisation
* Renal failure: serum creatinine >135 micromol/L
* Known liver disease with alkaline phosphatase or ALT >2x upper limit of reference range
* Bony fracture in past 3 months or Paget's disease of bone
* Secondary (central) hypothyroidism or hypopituitarism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55
Dates: Start 2003-04; Study Completion 2005-03

PRIMARY OUTCOMES:
Visual analog scales assessing wellbeing

SECONDARY OUTCOMES:
treatment satisfaction score
treatment preference
quality of life scores
cognitive function tests
clinical and biochemical markers of thyroid hormone action

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Charles Gairdner Hospital, Nedlands, Western Australia, Australia